CLINICAL TRIAL: NCT07116629
Title: A Community-Based Intervention To Address Health-Related Social Needs For Patients On LAI-PrEP
Brief Title: Catch A Vibe - 24-00864
Status: Not yet recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 24-00684
Record Dates: First submitted 2025-08-07; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Health-Related Social Needs
Keywords: LAI-PrEP; Community Partnerships; Health-Related Social Needs

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients on or initiating LAI-PrEP as part of standard of care: Quantitative HRSN surveys will be administered to Patient participants at enrollment, 4-, 8-, and 12-month visits to evaluate changes in HRSN, barriers/facilitators to resolving HRSN, and the impact of HRSN on LAI-PrEP persistence and retention in HIV care.
- Medical Staff who work with patients on LAI-PrEP: Survey will be administered to Medical Staff participants 6 months after enrollment of the first patient participant.
- CBO Partners who work with patients on LAI-PrEP linkage and addressing HRSN: Survey will be administered to community-based organization (CBO) Partner participants 6 months after enrollment of the first patient participant.
- Patients who decline LAI-PrEP as part of standard of care: Survey will be administered to Patients Who Decline LAI-PrEP to better understand why they declined LAI-PrEP.

SUMMARY:
This study evaluates a proposed community-based implementation strategy to scale up screening, identification, and intervention on Health-Related Social Needs (HRSN) among persons on Long-Acting Injectable Pre-exposure Prophylaxis (LAI-PrEP). To do so, (1) screening for HRSN will occur at provider visits every 4 months, (2) navigation and establishment of connections with community resources through collaboration with two established community-based organization (CBO) partners, and (3) development of a tracking system integrated into the Electronic Medical Record (EMR) for monitoring and assessment of referral outcomes.

ELIGIBILITY:
Inclusion Criteria:

For Patient participant group: In order to be eligible for participation in this study, an individual must meet all of the following criteria:

* 18 years of age or older
* Does not have HIV AND vulnerable for HIV infection per WHO, NHS, and CDC recommendations
* On or initiating LAI-PrEP as part of standard of care prior to study participation
* Identify as either a Black/Latine cisgender woman OR Black/Latine MSM OR Transgender or Nonbinary Individual
* Capacity and willingness to provide consent

For Medical Staff participant group: In order to be eligible for participation in this study, an individual must meet all of the following criteria:

* 18 years of age or older
* Works with patients who go to the Bellevue Pride Center
* Be employed at NYU Langone Health or NYC H+H/Bellevue as one of the following occupations

  * Physician
  * Clinical Pharmacist
  * Nurse
  * Medical Phlebotomist
  * Social Worker/Navigator
  * Community Health Worker
  * Medical Leader (i.e., director of services)

For CBO Partner participant group: In order to be eligible for participation in this study, an individual must meet all of the following criteria:

* 18 years of age or older
* Works with patients who go to the Bellevue Pride Center
* Be employed at one of the established CBOs
* Capacity and willingness to provide consent

For Patient Who Declines LAI-PrEP participant group: In order to be eligible for participation in this study, an individual must meet all of the following criteria:

* 18 years of age or older
* Declines LAI-PrEP as part of standard of care
* Capacity and willingness to provide consent

Exclusion Criteria:

For Patient participant group: An individual who meets any of the following criteria will be excluded from participation in this study:

* Less than 18 years old
* Known HIV seropositive status or test positive at screening
* Does not identify as one of the listed priority populations
* Not fluent in either English or Spanish
* Not interested in HIV PrEP
* Not willing to consent for study participation
* Does not reside within New York State
* Pregnant or planning to become pregnant at the time of consent.
* Without capacity to consent to participate in the study

For Medical Staff participant group: An individual who meets any of the following criteria will be excluded from participation in this study:

* Do not work with patients who go to the Bellevue Pride Center
* Is not employed at NYU Langone Health or NYC/H+H Bellevue as one of the following occupations

  * Physician
  * Clinical Pharmacist
  * Nurse
  * Medical Phlebotomist
  * Social Worker
  * Community Health Worker
  * Medical Leader (i.e., directors of services)

For CBO Partner participant group: An individual who meets any of the following criteria will be excluded from participation in this study:

• Does not work with patients who go to the Bellevue Pride Center

For Patient Who Declines LAI-PrEP participant group: An individual who meets any of the following criteria will be excluded from participation in this study:

* Less than 18 years old
* Interested in initiating LAI-PrEP as part of standard of care or on LAI-PrEP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There are multiple participant groups:
  * Patients on or initiating LAI-PrEP as part of standard of care
  * Medical Staff who work with patients on LAI-PrEP
  * CBO Partner who work with patients on LAI-PrEP
  * Patients who decline LAI-PrEP as part of standard of care
Sampling Method: Non-Probability Sample
Enrollment: 343 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Completion Rate of HRSN Screener | Baseline; Month 4; Month 8; Month 12

SECONDARY OUTCOMES:
Percentage of Participants who Identify Financial Insecurity as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Transportation as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Food Insecurity as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Legal Assistance as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Housing Insecurity and/or Homelessness as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Inadequate Housing as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Education as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Identify Employment as an HRSN | Baseline; Month 4; Month 8; Month 12
Percentage of Participants who Childcare Issues as an HRSN | Baseline; Month 4; Month 8; Month 12
PrEP Persistence | Baseline; Month 4; Month 8; Month 12
  Percentage of patients who remain on PrEP.
Retention in HIV Prevention Care | Baseline; Month 4; Month 8; Month 12
  Percentage of patients who are retained in HIV prevention care.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pitts, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYC Health + Hospitals/Bellevue, New York, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared. Requests should be directed to Robert.pitts@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose (individual participant data meta-analysis) will be granted access. Requests should be directed to Robert.pitts@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.